CLINICAL TRIAL: NCT02442921
Title: The Effect of Colchicine Treatment on the Progression of Proteinuria in Patients With Diabetic Nephropathy.
Brief Title: Colchicine for Diabetic Nephropathy Trial
Acronym: CDNT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: D-Cure, Israel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-2015-1560-SK-CTIL
Record Dates: First submitted 2015-04-30; First posted 2015-05-13 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine (Experimental): 20 patients will receive up to 2 mg of colchicine for 18 months
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): 20 patients will receive placebo for 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — up to 2mg of Colchicine daily
  Arms: Colchicine
Drug: Placebo — Daily placebo
  Arms: Placebo

SUMMARY:
Forty patients with diabetic nephropathy will be treated with colchicine up to 2 mg, or placebo, for 18 months. A follow up will be performed after 12 additional months. The primary outcome will be a significant reduction or stabilization of proteinuria during the 18 month treatment period.

DETAILED DESCRIPTION:
Diabetic nephropathy is the leading cause today for end stage renal failure in the western world. Multifactorial intervention in patients may slow the rate of albuminuria and renal injury; however several new drug trials have failed so far to significantly attenuate its progression. Several pathways are identified in the development of diabetic nephropathy, however, in recent years many researchers suspect that inflammatory pathways play central roles in the progression of diabetic neuropathy . There is compelling evidence that diabetes mellitus has an auto-inflammatory component with Nlrp3 inflammasome and interleukin -1 β activation. Colchicine is a relatively safe anti-inflammatory drug used to treat and reverse albuminuria in familial Mediterranean fever nephropathy, an auto-inflammatory disease. Data from one study demonstrated that colchicine diminished proteinuria and inflammation in experimental-diabetic animal models.

Working hypothesis and aims:

To assess whether colchicine reduces proteinuria in diabetic patients with diabetic neuropathy , despite maximal multi-factorial interventions (angiotensin-converting-enzyme inhibitors, tight glycemic and hypertensive control, lifestyle intervention, etc.).

Methods:

Forty patients with stable diabetes, and diabetic neuropathy with proteinuria of 0.5-6g/24 hours, despite standard treatment, will receive colchicine (n=20) or placebo (n=20) for 18 months. Urinary protein and creatinine clearance will be assessed three months before the study initiation, at baseline and every three months thereafter. Blood creatinine, complete blood count, creatine phosphokinase , liver function tests, fasting Glucose Test, HbA1c, and urine protein/creatinine ratio and diabetes mellitus treatment monitoring and follow-up will be performed every three months. Oral colchicine treatment will be initiated at 1mg per day, and increased gradually to 2 mg, if gastrointestinal or musculoskeletal disturbances are absent or tolerated. The participants will be called and evaluated a year after the end of treatment for all parameters mentioned. Statistical analysis will be performed by a statistician.

Expected results:

A significant reduction or stabilization of proteinuria during the 18 month treatment period, or at follow up at one year later.

Importance and Relevance to the call This study may define a new treatment for diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diabetes mellitus , age>18 years old, able to sign an informed consent.
2. Hemoglobin A1c in the range of 6-9%, stable for last year (0.5±)
3. Blood creatinine lower than 2 mg/dL.
4. Blood pressure lower than 140/90 mmHg on stable anti-hypertensive treatment for at least 3 months.
5. Treated with ACE or angiotensin II receptor blocker , unless contraindicated

Exclusion Criteria:

1. Malignancy or significant heart, lung or liver disease.
2. Any GI disease, inflammatory bowel disease , malnutrition ( BMI under 18 )
3. Psychiatric disease
4. Any muscle disease, history of rhabdomyolysis , myopathy or myositis.
5. Any disease causing renal injury/proteinuria apart from diabetes mellitus
6. Any inflammatory or autoimmune disease
7. Any infection during the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02-22 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of urinary protein excretion ( mg/24hrs) from baseline to 18 months. | From baseline to 18 months ( end of trial )

CONTACTS AND LOCATIONS:
Overall Officials: Shaye Kivity, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes